CLINICAL TRIAL: NCT03528031
Title: Habitual Diet and Avocado Trial
Acronym: HAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00047011
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2021-06

CONDITIONS: Intra-abdominal Fat; Metabolic Syndrome; High Cholesterol; Triglycerides High; Diet Habit; High Blood Sugar; Liver Fat; Dietary Modification; HDL Cholesterol, Low Serum; Cardiovascular Diseases; High Density Lipoprotein Deficiency; Low-density-lipoprotein-type; Cardiovascular Risk Factor; Diabetes
MeSH Terms: conditions — Metabolic Syndrome; Hypercholesterolemia; Hypertriglyceridemia; Feeding Behavior; Hyperglycemia; Fatty Liver; Hypoalphalipoproteinemias; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This clinical trial aims to assess the effect of providing one avocado per day on established parameters of health in comparison with a control group maintaining their habitual diets. Participants are pre-screened over the telephone initially to assess eligibility and likelihood of compliance. For those that remain eligible, additional screening is conducted at a study visit. Participants' eligibility is confirmed by the data entry system on the trial website when the Inclusion/Exclusion form is complete and entered. Randomization is performed automatically by the data entry system using a block design and stratified by site. Participants are randomly assigned to one of two equally sized groups. Neither participants nor staff will be blinded to intervention assignment. Both groups are instructed to continue to follow their habitual diet but the intervention group will receive one avocado per day. Participants are followed for outcomes for a six-month period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Daily Avocado (Experimental): Participants will follow their usual diet and lifestyle but also be provided with 1 avocado to consume per day for 6 months. To maximize compliance, participants will be provided with resources on how to choose, store and ripen avocados along with simple usage ideas. Specific nutrition guidance will not be provided. Participants will pick up fresh avocados every 2 weeks with minimal interaction with study personnel. Compliance visits will be conducted monthly.
  Interventions: Other: Intervention Daily Avocado
- Control Usual Diet and Lifestyle (No Intervention): Participants will be instructed to follow their usual diet and lifestyle. Participants will be allowed to consume up to 2 avocados per month, but avocado consumption will not be encouraged and no avocados will be provided. Compliance visits will be conducted monthly.

INTERVENTIONS:
Other: Intervention Daily Avocado — Participants follow their usual diet and lifestyle but also are provided with 1 avocado to consume per day for 6 months.
  Arms: Intervention Daily Avocado

SUMMARY:
The Habitual Diet and Avocado Trial will evaluate the effects of providing one avocado per day for recommended consumption over a 6 month period in a cohort of approximately 1000 free-living participants with increased waist circumference in comparison with a control group that will maintain their habitual diets. Participants will be recruited and screened at 4 clinics in 4 locations: Pennsylvania State University; Loma Linda University; UCLA, and Tufts University (250 per site).

DETAILED DESCRIPTION:
Preliminary evidence suggests that consumption of avocados can modulate body weight, food intake and markers of metabolic syndrome and may reduce visceral adiposity. Visceral adipose tissue is positively correlated with risk of cardiometabolic syndrome that predisposes to cardiovascular disease and diabetes. The Habitual Diet and Avocado Trial (HAT) aims to investigate an impactful outcome (visceral fat reduction) in a relevant population (Americans with an increased weight circumference) with a reasonable lifestyle modification (consumption of 1 avocado per day). HAT will evaluate the effect of providing one avocado per day for consumption over a 6 month period on established health parameters, including visceral adiposity, hepatic lipid content, markers of metabolic syndrome and high sensitivity C-reactive protein (hsCRP) when compared to a habitual diet. Blood specimens will be drawn and analyzed for fasting total cholesterol, triglyceride, HDL-C, glucose, insulin, hsCRP and RBC fatty acid profiles. Two non-contrast MRIs will be performed (at screening to assess eligibility and final participant visit 8 for randomized participants) to assess the volume of visceral adipose tissue and hepatic fat fraction. Four 24-hour dietary recalls will be conducted for study participants to capture dietary intake data. Questionnaires include the following: health and demographic including eating habits and physical activity; diet, food and avocado satisfaction (intervention group only); quality of life; and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Increased waist circumference defined as ≥35 inches for women, ≥40 inches for men
* At least 25 years old at screening
* Not currently eating more than 2 avocados per month (habitual intake in U.S.)

Exclusion Criteria:

* Does not eat avocados
* Sensitive / allergic to avocados
* Allergies to latex or oral allergy syndrome
* Not willing or unable to undergo MRI scans
* Unstable medical condition such as on dialysis for renal disease, cardiac, gastrointestinal, or hepatic disease, cancer (non-melanoma skin cancer >5 years ago acceptable, any cancer site >10yrs without recurrence).
* Pregnant, lactating, intention of pregnancy
* Lost or gained 10 lbs of body weight in last year
* Following restricted or weight loss dietary patterns
* Unstable anti-anxiety / anti-depressive / anti-psychotic medication use defined as dose change within last 6 months
* Oral steroid use within the last 6 months longer than 7 days
* Elevated alcohol intake (7+ drinks/week females; 14+ drinks/week males)
* Participation in another clinical intervention trial within 30 days of baseline
* PI judgment

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Visceral adiposity | Visit 1 (Screening, -2 to 0 weeks) and Visit 8 (26 weeks)
  Non-contrast MRI scans will be performed to assess the volume of visceral adipose tissue. The outcome will be pre-post difference, compare the estimated mean change from baseline to follow-up in the 2 randomized groups with all tests of group differences performed according to the intent to treat.

SECONDARY OUTCOMES:
Hepatic lipid content | Visit 1 (Screening, -2 to 0 weeks and Visit 8 (26 weeks)
  Non-contrast MRI scans will be performed to assess hepatic lipid content/hepatic fat fraction.
Metabolic syndrome markers (serum triglycerides, serum cholesterol, fasting serum glucose, fasting insulin) | Visit 2 (Baseline visit 0 weeks), Visit 5 (12 weeks), Visit 8 (26 weeks)
  Phlebotomy is performed after a minimum 8 hour fast. Specimens will be separated and aliquoted, and shipped for analysis to Tufts University site for: fasting total cholesterol, triglyceride, high density lipo-protein cholesterol (HDL-C), glucose and insulin. LDL will be calculated using the Friedewald equation unless fasting triglyceride levels are > 400 mg/dL in which case they will be measured using a direct LDL assay. There will be a comparison of the estimated mean change from baseline to follow-up with all tests of group differences performed according to intent to treat.
High-sensitivity C-reactive protein (hs-CRP) | Visit 2 (baseline/randomization, Week 0), Visit 5 (12 weeks), Visit 8 (26 weeks)
  C-reactive protein (CRP) is a protein that the liver makes when there is inflammation in the body. Also called a marker of inflammation and can be measured with the hs-CRP test. Inflamed arteries puts individuals at greater risk of heart disease, heart attack, stroke and peripheral arterial disease. A fasting sample will be obtained, shipped to and analyzed at Tufts University for hsCRP.
Red blood cell (RBC) monounsaturated fat/polyunsaturated fat (MUFA/PUFA) ratio | Visit 2 (Baseline/Randomization Visit, 0 weeks), Visit 5 (12 weeks), Visit 8 (26 weeks)
  Fasting RBC specimens shipped to Tufts University for analysis of RBC fatty acid profiles. The Fatty Acid Profile measures major fatty acids found in red blood cells.
Blood pressure | Visit 2 (baseline/randomization 0 weeks) Visit 3 (4 weeks), Visit 4 (8 weeks), Visit 5 (12 weeks), Visit 6 (16 weeks), Visit 7 (10 weeks), Visit 8 (26 weeks)
  Seated blood pressure will be measured at each visit (except the screening visit) utilizing automated devices as per a standardized protocol across all sites. Three measurements will be taken after a 5 minute rest period, 1 minute apart. The last two readings are averaged for analysis.
Weight | Visit 2 (baseline/randomization), Visit 5 (12 weeks) and Visit 8 (26 weeks-final)
  Participants will be weighed at all in-study visits using high quality digital scales commonly used in clinical practice and that are in good working order. Participants will be weighed in light street clothes without shoes. The same scale is used throughout the trial.
Waist circumference | Visit 1 (screening -2 to 0 weeks), Visit 2 (baseline/randomization 0 weeks), Visit 5 (12 weeks), Visit 8 (26 weeks)
  A measuring tape specifically designed for waist circumference (recommended brands include Gulick or Seca) will be used according to a standardized procedure outlined in the trial Manual of Procedures. Waist circumference will be used during screening to assess eligibility. Measurements will be taken against the skin at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Two measurements are obtained at each visit and averaged.
Diet, Food and Avocado Satisfaction | Visit 2 (baseline/randomization, 0 weeks), Visit 5 (12 weeks), Visit 8 (26 weeks)
  Questions regarding participant satisfaction with the diet and food intervention will be assessed by completing the Diet, Food and Avocado Satisfaction Questionnaire. The questionnaire will only be completed by participants randomized to consume one avocado a day. The questionnaire is completed within 24 hours of a clinic visit and can be self- or staff administered. It consists of 14 questions about eating and preparing avocados each having a 100 point Likert scale with responses of "Not at all" and "Extremely".
Quality of life RAND 36-Item Short Form Survey Instrument (SF-36) | Visit 2 (baseline), Visit 5 (12 weeks) and Visit 8 (26 weeks-final)
  All participants will complete the RAND (research and development) 36-Item Health Survey to assess 8 health concepts: physical functioning, bodily pain, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue and general health perceptions.All items are scored so that a high score defines more favorable health state. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100. Items in the same scale are averaged together to create 8 scale scores. Items that are left blank are not taken into account when calculating scale scores.
Quality of Life RAND 20-Item Short Form Survey (SF-20) | Visit 3 (4 weeks), Vist 4 (8 weeks) Visit 6 (16 weeks), Visit 7 (20 weeks)
  The 20-item Short Form Health Survey (SF-20) was designed to reduce respondent burden while achieving minimum standards of precision for purposes of group comparisons involving multiple health dimensions. It includes 7 items to assess physical functioning, 2 items on role functioning, 1 social functioning survey item, 5 items to assess mental health, 4 items on current health perceptions and 1 item on pain. Participants in the control group will complete the RAND 20-Item Short Form Survey.
Sleep quality | Visit 2 (baseline), Visit 5 (12 weeks) and Visit 8 (26 weeks-final)
  All participants will complete the Pittsburgh Sleep Quality Index questionnaire (PSQI) which is a self-rated questionnaire that assesses sleep quality and disturbances over a 1-month time time interval. 19 individual items generate seven "component" scores: subjective sleep quality; sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction. The sum of scores for the 7 components yield one global score.
24-hour diet recall | Visit 1 (screening, -2 to 0 weeks), Visit 4 (8 weeks), visit 6 (16 weeks), Visit 8 (26 weeks)
  Four 24-hour dietary recalls will be conducted for each study participant during the course of the study. The goal for the 3 intra-study recalls is to capture intake data for 2 weekdays and 1 weekend day for each participant. The recalls are collected and analyzed using Nutrition Data System for Research (NDSR) software Vs 2017. The Loma Linda University site and Tufts University will be responsible for collecting 50% each of the 24 hour recalls across all study sites. They will follow a standardized manual of procedures for dietary data collection and dietary data management. Outcome data from NDSR will include daily estimated energy and nutrient intake, as well as food, food group and dietary supplement data.

CONTACTS AND LOCATIONS:
Overall Officials: David Reboussin, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (4):
- United States (4):
  - Loma Linda University, Loma Linda, California
  - University of California Los Angles (UCLA), Los Angeles, California
  - Tufts University, Boston, Massachusetts
  - Pennysylvania State University, University Park, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Investigators may wish to perform ancillary studies using the HAT population, samples or other collected data. All ancillary studies must be approved by the HAT Steering Committee before being allowed access to study participant, samples or the database. De-identified individual participant data for all primary and secondary outcome measures will be made available to participating sites and for at the end of the study and for public use databases.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed by the Steering Committee. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Result] Berryman CE, West SG, Fleming JA, Bordi PL, Kris-Etherton PM. Effects of daily almond consumption on cardiometabolic risk and abdominal adiposity in healthy adults with elevated LDL-cholesterol: a randomized controlled trial. J Am Heart Assoc. 2015 Jan 5;4(1):e000993. doi: 10.1161/JAHA.114.000993. PMID 25559009
- [Result] Bertoli S, Leone A, Vignati L, Bedogni G, Martinez-Gonzalez MA, Bes-Rastrollo M, Spadafranca A, Vanzulli A, Battezzati A. Adherence to the Mediterranean diet is inversely associated with visceral abdominal tissue in Caucasian subjects. Clin Nutr. 2015 Dec;34(6):1266-72. doi: 10.1016/j.clnu.2015.10.003. Epub 2015 Oct 20. PMID 26499033
- [Result] Cespedes Feliciano EM, Tinker L, Manson JE, Allison M, Rohan T, Zaslavsky O, Waring ME, Asao K, Garcia L, Rosal M, Neuhouser ML. Change in Dietary Patterns and Change in Waist Circumference and DXA Trunk Fat Among Postmenopausal Women. Obesity (Silver Spring). 2016 Oct;24(10):2176-84. doi: 10.1002/oby.21589. Epub 2016 Aug 22. PMID 27548405
- [Result] Dhillon J, Tan SY, Mattes RD. Almond Consumption during Energy Restriction Lowers Truncal Fat and Blood Pressure in Compliant Overweight or Obese Adults. J Nutr. 2016 Dec;146(12):2513-2519. doi: 10.3945/jn.116.238444. Epub 2016 Nov 2. PMID 27807041
- [Result] Estruch R, Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ruiz-Gutierrez V, Covas MI, Fiol M, Gomez-Gracia E, Lopez-Sabater MC, Vinyoles E, Aros F, Conde M, Lahoz C, Lapetra J, Saez G, Ros E; PREDIMED Study Investigators. Effects of a Mediterranean-style diet on cardiovascular risk factors: a randomized trial. Ann Intern Med. 2006 Jul 4;145(1):1-11. doi: 10.7326/0003-4819-145-1-200607040-00004. PMID 16818923
- [Result] Gower BA, Goss AM. A lower-carbohydrate, higher-fat diet reduces abdominal and intermuscular fat and increases insulin sensitivity in adults at risk of type 2 diabetes. J Nutr. 2015 Jan;145(1):177S-83S. doi: 10.3945/jn.114.195065. Epub 2014 Dec 3. PMID 25527677
- [Result] Paniagua JA, Gallego de la Sacristana A, Romero I, Vidal-Puig A, Latre JM, Sanchez E, Perez-Martinez P, Lopez-Miranda J, Perez-Jimenez F. Monounsaturated fat-rich diet prevents central body fat distribution and decreases postprandial adiponectin expression induced by a carbohydrate-rich diet in insulin-resistant subjects. Diabetes Care. 2007 Jul;30(7):1717-23. doi: 10.2337/dc06-2220. Epub 2007 Mar 23. PMID 17384344
- [Result] Ross R, Rissanen J, Pedwell H, Clifford J, Shragge P. Influence of diet and exercise on skeletal muscle and visceral adipose tissue in men. J Appl Physiol (1985). 1996 Dec;81(6):2445-55. doi: 10.1152/jappl.1996.81.6.2445. PMID 9018491
- [Result] National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. Circulation. 2002 Dec 17;106(25):3143-421. No abstract available. PMID 12485966
- [Result] Wien M, Haddad E, Oda K, Sabate J. A randomized 3x3 crossover study to evaluate the effect of Hass avocado intake on post-ingestive satiety, glucose and insulin levels, and subsequent energy intake in overweight adults. Nutr J. 2013 Nov 27;12:155. doi: 10.1186/1475-2891-12-155. PMID 24279738
- [Result] O'Neil, et al. Avocado consumption by adults is associated with better nutrient intake, diet quality and some measures of adiposity: NHANES Survey, 2001-2012. Int Med Rev In press.
- [Derived] Damani JJ, Kris-Etherton PM, Lichtenstein AH, Matthan NR, Sabate J, Li Z, Reboussin D, Petersen KS. Effect of Daily Avocado Intake on Cardiovascular Health Assessed by Life's Essential 8: An Ancillary Study of HAT, a Randomized Controlled Trial. J Am Heart Assoc. 2025 Mar 4;14(5):e039130. doi: 10.1161/JAHA.124.039130. Epub 2025 Feb 19. PMID 39968784
- [Derived] Clarke AE, LeBeau KS, Oda K, Segovia-Siapco G, Paalani M, Reboussin DM, Lichtenstein AH, Rajaram S, Sabate J. The Effect of Daily Avocado Intake on Food and Nutrient Displacement in a Free-Living Population with Abdominal Obesity. Curr Dev Nutr. 2024 Aug 27;8(10):104451. doi: 10.1016/j.cdnut.2024.104451. eCollection 2024 Oct. PMID 39886351
- [Derived] Yang J, Lei OK, Bhute S, Kris-Etherton PM, Lichtenstein AH, Matthan NR, Petersen KS, Sabate J, Reboussin DM, Lovato L, Vitolins MZ, Rajaram S, Jacobs JP, Huang J, Taw M, Yang S, Li Z. Impact of daily avocado consumption on gut microbiota in adults with abdominal obesity: an ancillary study of HAT, a randomized controlled trial. Food Funct. 2025 Jan 2;16(1):168-180. doi: 10.1039/d4fo03806a. PMID 39641169
- [Derived] Matthan NR, Lovato L, Petersen KS, Kris-Etherton PM, Sabate J, Rajaram S, Li Z, Reboussin DM, Lichtenstein AH. Effect of daily avocado consumption for 6 mo compared with habitual diet on red blood cell fatty acid profiles and association with cardiometabolic risk factors in individuals with abdominal obesity: a randomized trial. Am J Clin Nutr. 2024 Oct;120(4):794-803. doi: 10.1016/j.ajcnut.2024.08.002. Epub 2024 Aug 10. PMID 39128497
- [Derived] Davis KM, Petersen KS, Matthan NR, Legro RS, Kris-Etherton PM. Effect of Incorporating 1 Avocado per Day Versus Habitual Diet on Vascular Function in Adults With Abdominal Obesity: An Ancillary Study of HAT, a Randomized Controlled Trial. J Am Heart Assoc. 2024 May 21;13(10):e030497. doi: 10.1161/JAHA.123.030497. Epub 2024 May 10. PMID 38726886
- [Derived] Petersen KS, Smith S, Lichtenstein AH, Matthan NR, Li Z, Sabate J, Rajaram S, Segovia-Siapco G, Reboussin DM, Kris-Etherton PM. One Avocado per Day as Part of Usual Intake Improves Diet Quality: Exploratory Results from a Randomized Controlled Trial. Curr Dev Nutr. 2024 Jan 11;8(2):102079. doi: 10.1016/j.cdnut.2024.102079. eCollection 2024 Feb. PMID 38375072
- [Derived] Lichtenstein AH, Kris-Etherton PM, Petersen KS, Matthan NR, Barnes S, Vitolins MZ, Li Z, Sabate J, Rajaram S, Chowdhury S, Davis KM, Galluccio J, Gilhooly CH, Legro RS, Li J, Lovato L, Perdue LH, Petty G, Rasmussen AM, Segovia-Siapco G, Sirirat R, Sun A, Reboussin DM. Effect of Incorporating 1 Avocado Per Day Versus Habitual Diet on Visceral Adiposity: A Randomized Trial. J Am Heart Assoc. 2022 Jul 19;11(14):e025657. doi: 10.1161/JAHA.122.025657. Epub 2022 Jul 5. PMID 35861827

DOCUMENTS (1):
  • Informed Consent Form (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/31/NCT03528031/ICF_000.pdf